CLINICAL TRIAL: NCT06123533
Title: An Exploratory Study to Understand Women's Values of Management of a Positive Human Papillomavirus (HPV) Test From the Cervical Screening Programme
Brief Title: Understanding Women's Values in Managing Human Papillomavirus (HPV)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2-039-23
Record Dates: First submitted 2023-10-31; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Human Papilloma Virus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — There is no intervention.

SUMMARY:
Almost all cervical cancers are caused by infection with a high-risk (hr) HPV. In March 2020, the Scottish Cervical Screening programme changed from a test to look for abnormal cervical cells caused by hr-HPV to a test that looks for infection with hr-HPV itself. If an HPV infection persists, there is an increased risk of a pre-cancer or cancer of the cervix developing in the future. The cervical screening programme aims to detect and treat pre-cancers, so they don't progress to cancer of the cervix.

Most HPV infections do not cause symptoms and will clear on their own. There are no active treatments available currently. Following a positive hr-HPV result, by waiting and repeating the HPV test after 12 months, it is known that 60% of infections clear in that year and more will clear each year after. Some women are anxious when they find out that they have an HPV infection, and some will look to see if there are any treatments available.

Several private organisations are offering HPV treatments which are not approved for clinical use yet. These may, or may not, help clear up HPV more quickly or more often.

This study is designed to help us to know and understand whether women have considered treatments, which benefits or risks of such treatments they value, and which factors influence these decisions. The study will also seek to determine participants' willingness to pay for such treatments and will also help to facilitate discussions between clinicians and patients.

DETAILED DESCRIPTION:
A scoping review was conducted to determine the background information and evidence available with regards to treatment of persistent human papillomavirus (HPV) in women. This scoping review, which will become a systematic review, evidenced that there was a knowledge gap on how to manage persistent HPV. Several different treatment options were identified, with some studies being conducted as randomised controlled trials and some being conducted as cohort studies.

In March 2020, the Scottish Cervical Screening programme changed from cervical cytology test (test of disease; testing of cells taken by a brush from the cervix and analysed under a microscope) to testing for high-risk HPV (a test of risk). If an HPV infection persists, there is an increased risk of having precancer or cancer of the cervix in the future.

Informing women that they have a viral infection which can result in cancer has in effect created a 'new disease' as women would not have been aware of this infection. Most HPV infections do not cause symptoms and there are no active treatments available in the NHS. This has created concerns for some women who may want to find a treatment and feel that surveillance, where 60% of infections should regress is 'doing nothing.'

Several private organisations are offering HPV treatments which are not available in the NHS, and which may help clear up HPV including HPV vaccination, and probiotics and vaginal gels. This proposal will take steps towards understanding an unmet need among women who have high-risk HPV and who are on early repeat HPV testing. It will seek to understand whether women have considered treatments, which benefits, or risks of such treatments are valued, and which factors influence these decisions as a health economics study.

Although these treatments require further evidence and development prior to being adopted as options for patient care, conducting this research will provide valuable insights into what women value. The profiles of the different treatments vary significantly and understanding patient preferences will help guide prioritisation. Understanding initially how women feel about their HPV diagnosis and the available treatments will be important to design a pilot discrete choice experiment (DCE) and usable DCE to understand, in quantitative terms, what women seek, prioritise and are willing to pay for in their care for HPV.

This study is being performed to provide valuable insights to conduct a DCE. The results of the participant interviews and the DCE will be highly useful to help inform policy, guidelines and clinical recommendations for the management of women with persistent HPV.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, English speaking, female patients aged 25-64 years
* Women with cervical high risk HPV infection
* Normal colposcopy, or, if cytological or histological changes present at colposcopy, a diagnosis of borderline nuclear abnormalities, low grade dyskaryosis or CIN1 only

Exclusion Criteria:

* Cytological or histological diagnosis of CIN2+, high grade dyskaryosis, or cervical cancer at colposcopy
* Planned treatments that involve surgical excision e.g. LEEP, LLETZ, conisation or ablation of cervix
* Chronic immunosuppression
* Limited English language proficiency

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be identified through their cervical screening record on Scottish Cervical Call Recall System (SCCRS) records at the Women's Day Clinic (colposcopy clinic) in NHS Grampian.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-06 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
% of participants who feel certain key factors of care are important to them in making choices about how to manage their HPV diagnosis. | March 2024
  Participants will be asked about a number of factors and their opinions on how they influence their treatment decisions, including price, mode of treatment, frequency of treatment and duration of treatment. Interview transcripts will be analysed to determine themes through thematic analysis. This will allow the investigators to understand what is important to participants. This information is required to create a pilot DCE, to further understand the wants and needs of those with persistent HPV.

IPD SHARING:
Plan to Share IPD: No